CLINICAL TRIAL: NCT04006015
Title: Activity, Balance and COPD: An Exploratory Study of Physical Activity and Balance in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Activity, Balance and COPD (ABCOPD)
Acronym: ABCOPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS Project ID: 258399
Record Dates: First submitted 2019-06-24; First posted 2019-07-02 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Main study group: 31 people with COPD and 31 controls in the main study group.
  Interventions: Other: No intervention being delivered.
- six-minute walk substudy: We will aim to have 40 participants participating in the 6 minute walk sub-study.
  Interventions: Other: No intervention being delivered.
- Qualitative dance substudy: We will aim for 20 participants.
  Interventions: Other: No intervention being delivered.

INTERVENTIONS:
Other: No intervention being delivered. — No interventions are being delivered.

SUMMARY:
This research project incorporates a series of studies to investigate the relationship between physical performance (e.g. tests of strength, balance and walking distance) and physical activity (activity measured in day to day life) in people with COPD and other chronic lung diseases.

DETAILED DESCRIPTION:
The research project incorporates the following components:

Study 1) A prospective, observational study, to assess the relationship between a comprehensive set of measures of walking ability, strength and balance, and daily physical activity in people with chronic lung disease. Patients will attend a single assessment session to evaluate physical capacity. They will also wear a physical activity monitor for a week following completing these tests to assess physical activity and aspects of physical performance. Participants will also be invited to return two months later to provide evidence about the repeatability of measurements.

Study 2) A parallel study comparing assessment of performance during six-minute walk tests by an observer to a semi-automated assessment using an activity monitor worn by the patient. This will involve a single visit and be carried out during walking tests carried out as part of routine clinical care.

Study 3) A qualitative study to investigate experiences and perceptions of participants of dance groups for people with chronic lung disease, as a novel form of physical activity. This will be used to inform the design of subsequent trials of dance interventions for chronic lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults with stable chronic lung disease
* Able to understand instructions.
* Age and sex matched healthy controls.

Exclusion Criteria:

* For the main study, the presence of other comorbidities causing a significant reduction in mobility (for example stroke with neurological deficits, severe arthritis, significant peripheral neuropathy, significant visual impairment, dementia etc.).
* exacerbation of lung disease within the last 2 months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with stable chronic lung disease.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Free-living gait stability as assessed by activity monitor | 7 days.
  The free-living gait stability parameters derived from the fixed body sensor worn during activity monitoring at home.

SECONDARY OUTCOMES:
Physical activity assessed by step count using activity monitor | 7 days.
  Physical activity assessed using step count (number of steps), as assessed using the activity monitor at home (McRoberts MoveMonitor).
Clinical balance assessment | Assessed during single clinical assessement at baseline.
  Assessed using the miniBESTest in clinical setting.
Physical performance assessment | Assessed during single clinical assessment at baseline.
  Assessed using the Short Physical Performance Battery (SPPB) in clinical setting.
Balance confidence | Assessed during a single clinical assessment at baseline.
  Assessed using the Activities-specific Balance Confidence (ABC) scale. This is a self completed measure of balance confidence during common activities of daily living. It includes 16 questions which participant give a percentage confidence response with 0% being not confident at all and 100% being completely confident. There is also a total score out from 0% (least confident) to 100% (most confident) for overall balance confidence, which average created by combining the scores given for the separate questions.
Walking distance in metres | Assessed during a single clinical assessment at baseline.
  Assessed using the six-minute walk test in clinical setting.
Patient experience as assessed by semi-structured interviews | 1 hour.
  The patients experience assessed by semi-structured interviews in focus group.
Physical Activity: Movement intensity (in average body acceleration (g) during activity) | 7 days.
  Movement intensity measurement is assessed using the fixed body sensor worn during activity monitoring at home.
Physical activity: types of activity (time in minutes spent standing, walking, lying, sitting, cycling, running) assessed with activity monitor. | 7 days.
  Types of activity (time measured in minutes spent standing, walking, lying, sitting, cycling, running) is assessed using the fixed body sensor worn during activity monitoring at home.
Timed Up and Go (TUG) | Assessed during a single clinical assessment at baseline.
  Time in seconds to complete the standard TUG protocol
Functional reach test | Assessed during a single clinical assessment at baseline.
  Assessed using standard functional reach protocol

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hopkinson, PhD, Principal Investigator — Imperial College London
Locations (1):
- National Heart and Lung Institute, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Philip KEJ, Lewis A, Williams S, Buttery SC, Polkey MI, Man W, Fancourt D, Hopkinson NS. Dance for people with chronic respiratory disease: a qualitative study. BMJ Open. 2020 Oct 13;10(10):e038719. doi: 10.1136/bmjopen-2020-038719. PMID 33051234